CLINICAL TRIAL: NCT02699164
Title: Lumbal Disk Herniasyonunda farklı Tedavi yöntemlerinin etkinliğinin karşılaştırılması
Brief Title: Remission of Lumbar Disc Herniation by Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Research asisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GO14-265
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Lumbar Disc Herniation
Keywords: non surgical spinal decompression therapy; deep friction massage; exercise
MeSH Terms: conditions — Intervertebral Disc Displacement; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- combine group (Experimental): Conventional physiotherapy applied 15 sessions of treatment. In addition to conventional physiotherapy non-surgical spinal decompression therapy applied.
  First 10 sessions of treatment non-surgical decompression therapy applied and last 5 sessions spinal stabilization exercise applied.
  Interventions: Device: DRX 9000, Axiom Worldwide, Tampa, Florida; Other: physiotherapy; Other: spinal stabilization exercise
- conventional physiotherapy (Experimental): conventional physiotherapy applied 15 sessions of treatment. Conventional physiotherapy consisted hotpack, Transcutaneal Electric Nerve Stimulation(TENS) and Ultrasound Currents. Spinal stabilization exercises applied last five sessions of therapy.
  Interventions: Other: physiotherapy; Other: spinal stabilization exercise

INTERVENTIONS:
Device: DRX 9000, Axiom Worldwide, Tampa, Florida — non-surgical spinal decompression therapy consist 18 traction cycles. Traction force applied herniation levels according to Magnetic Resonance Imaging (MRI).
  Arms: combine group
Other: physiotherapy — electrotherapy was used. electrotherapy consisted of 20 minutes of hot-pack, 20 minutes of TENS and 5 minutes of ultrasound.
Other: spinal stabilization exercise — spinal stabilization exercises started elementary exercises. According to patient tolerance, exercise program reestablished.

SUMMARY:
This study was conducted with the aim of determining whether or not Non surgical spinal decompression therapy was effective in remission of herniation, decreasing pain and improving functional status.

DETAILED DESCRIPTION:
Both groups received combination of electrotherapy, deep friction massage and stabilization exercise for fifteen session.

Combine group received non surgical spinal decompression therapy (NSDT) different from conventional physiotherapy group. Numeric Analog Scale, Straight leg raise (SLR) test, Oswestry Disability Index (ODI) were applied at baseline and after treatment. Disc height and herniation thickness were measured on Magnetic Resonance Imagination (MRI) which performed at baseline and three months after therapy.

ELIGIBILITY:
Inclusion Criteria:

diagnosed as lumbar disc herniation suffering from low back pain at least 8 weeks

Exclusion Criteria:

undergone any spinal surgery clinical diagnosis of osteoporosis clinical diagnosis of scoliosis and spondylolisthesis any neurological disease causes sensorial loss

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
herniation thickness | change from baseline in herniation thickness and disc height at three months
  herniation thickness were measured on MRI.

SECONDARY OUTCOMES:
function | up to 3 months
  Oswestry Disability Index was used.Oswestry Disability Index used to assess the changes in function and disability levels. Scores range from 0 to 100.
  scores between 0 and 20 described as "minimal disability", scores between 21and 40 described as "moderate disability",scores between 41and 60 described as "severe disability",scores between 61 and 80 described as "crippled" and scores between 81 and 100 described as " bed bounded"
mobility | up to 3 months
  straight leg raise test was used. Pain free angle of straight leg raise was measured with goniometer.
pain severity | change form baseline in pain severity at 15 sessions of treatment
  numeric analog scale was used. "0" described no pain, "10" described "unbearable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Principal Investigator — Hacettepe University; Nevin Ergun, Proff, Principal Investigator — Hacettepe University; Mehmet Yorubulut, MD, Principal Investigator — Acıbadem Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundon K, Bolton K. Structure and function of the lumbar intervertebral disk in health, aging, and pathologic conditions. J Orthop Sports Phys Ther. 2001 Jun;31(6):291-303; discussion 304-6. doi: 10.2519/jospt.2001.31.6.291. PMID 11411624
- [Result] Apfel CC, Cakmakkaya OS, Martin W, Richmond C, Macario A, George E, Schaefer M, Pergolizzi JV. Restoration of disk height through non-surgical spinal decompression is associated with decreased discogenic low back pain: a retrospective cohort study. BMC Musculoskelet Disord. 2010 Jul 8;11:155. doi: 10.1186/1471-2474-11-155. PMID 20615252
- [Result] Schoenfeld AJ, Weiner BK. Treatment of lumbar disc herniation: Evidence-based practice. Int J Gen Med. 2010 Jul 21;3:209-14. doi: 10.2147/ijgm.s12270. PMID 20689695
- [Result] Lurie JD, Tosteson AN, Tosteson TD, Carragee E, Carrino JA, Kaiser J, Sequeiros RT, Lecomte AR, Grove MR, Blood EA, Pearson LH, Herzog R, Weinstein JN. Reliability of magnetic resonance imaging readings for lumbar disc herniation in the Spine Patient Outcomes Research Trial (SPORT). Spine (Phila Pa 1976). 2008 Apr 20;33(9):991-8. doi: 10.1097/BRS.0b013e31816c8379. PMID 18427321
- [Result] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Hanscom B, Skinner JS, Abdu WA, Hilibrand AS, Boden SD, Deyo RA. Surgical vs nonoperative treatment for lumbar disk herniation: the Spine Patient Outcomes Research Trial (SPORT): a randomized trial. JAMA. 2006 Nov 22;296(20):2441-50. doi: 10.1001/jama.296.20.2441. PMID 17119140
- [Result] Romanowski M, Romanowska J, Grzeskowiak M. A comparison of the effects of deep tissue massage and therapeutic massage on chronic low back pain. Stud Health Technol Inform. 2012;176:411-4. PMID 22744541
- [Result] Hahne AJ, Ford JJ, Hinman RS, Taylor NF, Surkitt LD, Walters AG, McMeeken JM. Outcomes and adverse events from physiotherapy functional restoration for lumbar disc herniation with associated radiculopathy. Disabil Rehabil. 2011;33(17-18):1537-47. doi: 10.3109/09638288.2010.533814. Epub 2010 Nov 20. PMID 21091049
- [Result] Choi J, Lee S, Hwangbo G. Influences of spinal decompression therapy and general traction therapy on the pain, disability, and straight leg raising of patients with intervertebral disc herniation. J Phys Ther Sci. 2015 Feb;27(2):481-3. doi: 10.1589/jpts.27.481. Epub 2015 Feb 17. PMID 25729196